CLINICAL TRIAL: NCT04540172
Title: Music Therapy and Progressive Muscle Relaxation Exercise
Brief Title: The Effect of Music Therapy and Progressive Muscle Relaxation Exercise on Anxiety Before the First Clinical Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Demet İnangil, PhD, Asistant Professor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 46418926
Record Dates: First submitted 2020-09-04; First posted 2020-09-07 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Anxiety; Stress
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Therapy (Experimental): music therapy was applied in the practice room. Environmental noise was reduced as much as possible; the room was dimly lit. The students were asked to close their eyes after sitting comfortably in a chair and focus on the music by asking them to imagine a different memory and place that would relax them instead of the thoughts that occupied their minds. The music was played through a portable computer for 15 minutes under the supervision of the researchers using an mp3 player program on the computer.
  Interventions: Behavioral: Music Therapy
- Progressive Muscle Relaxation Exercise (Experimental): In this study, the steps of applying progressive muscle relaxation exercises were created with the guidance of the "Relaxation Exercises " materials of the Turkish Psychological Association. Warning messages were hung on the door of the room, environmental noise was reduced as much as possible, and the room was provided with dim lighting. The students were asked to close their eyes and breathe deeply after sitting comfortably in a chair. After taking two deep breaths, they were told to dangle their arms and relax as much as possible. The hands, shoulders, neck, chest, abdomen, hips, legs, feet, toes, and facial muscles were made to relax while they breathed and relaxed while exhaling. They were asked to store the experience into their memories thoroughly so that they could recall this feeling for comfort during the day.
  Interventions: Behavioral: Progressive Muscle Relaxation Exercise
- Control (No Intervention): No additional method was applied in the control group.

INTERVENTIONS:
Behavioral: Music Therapy — "Mahur tune," one of the nonverbal instruments of the Traditional Turkish Music Authorities, was selected for the study with the opinion of a music therapy specialist.
  Arms: Music Therapy
Behavioral: Progressive Muscle Relaxation Exercise — In this study, the steps of applying progressive muscle relaxation exercise were created with the guidance of the "Relaxation Exercises " materials of the Turkish Psychological Association.
  Arms: Progressive Muscle Relaxation Exercise

SUMMARY:
This study was carried out to evaluate the effect of music therapy and progressive muscle relaxation exercise on the state and trait anxiety levels before their first clinical practice in nursing students.

DETAILED DESCRIPTION:
This randomized controlled experimental study sample consisted of 86 nursing students who will be firstly applied to clinical practice. The students were randomly assigned to music (n=30), exercise (n=28), and control (n=28) groups. The data of the study were collected with Student Information Form and State-Trait Anxiety Scale. The music therapy intervention was applied to the experimental groups three times a week for the first 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years or older,
* being enrolled in the Nursing Fundamentals theoretical course,
* participating fully in the attempts being applied in the study,
* volunteering to participate in the study.

Exclusion Criteria:

* be graduating from Health Vocational High School
* not being in the field of application determined on the first clinical application day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Anxiety | Change from baseline in 1 week
  The level of Anxiety was evaluated with the State-Trait Anxiety Inventory (STAI). STAI consists of 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (None" (1), "A little" (2), "Very" (3), and "Completely" (4). Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Merdiye Şendir, PhD, Study Chair — Saglik Bilimleri University
Locations (1):
- Demet İnangil, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dehghan-Nayeri N, Adib-Hajbaghery M. Effects of progressive relaxation on anxiety and quality of life in female students: a non-randomized controlled trial. Complement Ther Med. 2011 Aug;19(4):194-200. doi: 10.1016/j.ctim.2011.06.002. Epub 2011 Jul 12. PMID 21827933
- [Background] Chen Y, Yang X, Wang L, Zhang X. A randomized controlled trial of the effects of brief mindfulness meditation on anxiety symptoms and systolic blood pressure in Chinese nursing students. Nurse Educ Today. 2013 Oct;33(10):1166-72. doi: 10.1016/j.nedt.2012.11.014. Epub 2012 Dec 20. PMID 23260618
- [Derived] Inangil D, Sendir M, Kabuk A, Turkoglu I. The Effect of Music Therapy and Progressive Muscle Relaxation Exercise on Anxiety Before the First Clinical Practice in Nursing Students: A Randomized Controlled Study. Florence Nightingale J Nurs. 2020 Oct 26;28(3):341-349. doi: 10.5152/FNJN.2020.19075. eCollection 2020 Oct. PMID 34263213